CLINICAL TRIAL: NCT03871153
Title: A Phase II Study of Concurrent Chemoradiation Plus Durvalumab (MEDI4736) Followed by Surgery Followed by Adjuvant Durvalumab (MEDI4736) in Medically Operable Patients With Surgically Resectable Stage III (N2) Non-Small Cell Lung Cancer
Brief Title: Chemoradiation Plus Durvalumab Followed by Surgery Followed by Adjuvant Durvalumab in Patients With Surgically Resectable Stage III (N2) Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decided to halt study due to low accrual.
Sponsor: Greg Durm, MD (Other)
Collaborators: AstraZeneca (Industry); Indiana University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Greg Durm, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCRN LUN17-321
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Non Small Cell Lung Cancer; Stage III Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Cisplatin; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other): Neoadjuvant chemotherapy(Durvalumab, Paclitaxel, Carboplatin), radiation and immunotherapy (durvalumab) followed by surgical resection followed by adjuvant immunotherapy (durvalumab)
  Interventions: Device: Durvalumab; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Radiation; Procedure: Surgical Resection

INTERVENTIONS:
Device: Durvalumab — Neoadjuvant Durvalumab 750 mg IV on Days 1, 15 and 29
  Adjuvant Durvalumab 12 weeks after undergoing surgical resection 1,500 mg IV on Day 1
  Other Names: Imfinzi
Drug: Paclitaxel — Paclitaxel 45 mg/m2 IV Days 1, 8, 15, 22, 29 and +/- 36
  Other Names: Taxol
Drug: Carboplatin — Carboplatin AUC of 2 IV Days 1, 8, 15, 22, 29 +/- 36
  Other Names: Platinol
Radiation: Radiation — 1.8-2.0 Gy per day (5 days/week) for a total of 45-61.2 Gy over 5-6 weeks. Treatment will be delivered using IMRT or 3DCRT using typically 6-10MV photons. Proton therapy is also allowed. 4D simulation and appropriate IGRT are encouraged. Radiation therapy must begin within one week of the first day of chemotherapy (or vice versa).
Procedure: Surgical Resection — Patients will undergo repeat imaging between 4 and 12 weeks after completing neoadjuvant therapy. Those without evidence of progressive disease and found to be a surgical candidate by a thoracic surgeon will undergo surgical resection between 4 and 12 weeks after neoadjuvant therapy.

SUMMARY:
This is an open label, multi-institutional, single arm Phase II trial. All patients will be treated with Carboplatin, Paclitaxel, Durvalumab and Radiation. All patients with non-PD after induction therapy who remain surgical candidates will undergo surgical resection 4-12 weeks following induction therapy.

After surgical resection, all patients who remain eligible will be treated with adjuvant Durvalumab every 4 weeks for 6 cycles beginning 4-12 weeks after surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0 or 1 within 28 days prior to registration.
* Histological or cytological confirmation of NSCLC (Adenocarcinoma, Squamous Cell Carcinoma, Large Cell Carcinoma). A pathology report (from the last 6 months) confirming the diagnosis of NSCLC must be obtained and reviewed by the treating physician prior to registration to study.
* Must have resectable and medically operable stage III (N2) NSCLC with clinical or biopsy-proven N2 disease. If patients have clinical N2 disease they need to be biopsy-proven (with EBUS or mediastinoscopy) during screening and have confirmed prior to study enrollment). Subjects must be considered resectable and medically operable based on the judgment of the treating physician. Stage III (N2) defined as per the 7th edition of the TNM staging system (T1a, T1b, T1c, T2a, T2b, T3, or T4)N2M0.
* Individuals cannot have contralateral neck or contralateral mediastinum nodal involvement.
* Subjects must have a life expectancy of at least 12 weeks to qualify.
* Individuals must not have distant metastasis, defined as M0 in the TMN staging system.
* Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 28 days prior to registration.

  * Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3
  * Hemoglobin (Hgb) ≥ 9 g/dL (may be transfused)
  * Platelets ≥100,000/mcl
  * Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 x upper limit of normal (ULN) OR ≥ 40 mL/min for subjects with creatinine levels >1.5 x institutional ULN
  * Bilirubin ≤ 1.5 × ULN OR Direct bilirubin of ≤ ULN for subjects with total bilirubin levels of >1.5x ULN
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN if no liver metastases

    ≤ 5 x ULN if liver metastases present
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN if no liver metastases ≤ 5 x ULN if liver metastases present
* All CT or PET imaging studies must be completed within 6 weeks (42 days) prior to registration.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to registration. NOTE: Women are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 62 must have a documented serum follicle stimulating hormone (FSH) level greater than 40 mIU/mL.
* Women of childbearing potential must be willing to abstain from heterosexual activity or use an effective method of contraception from the time of informed consent until 90 days after treatment discontinuation.
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving study drug and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 90 days after the last dose of investigational product.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* History of a major surgical procedure (as defined by investigator) within 28 days prior to the first dose of study drug. NOTE: Local surgery for isolated lesions for palliative intent is acceptable.
* History of another primary malignancy except for a) malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study drug, b) adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, c) adequately treated carcinoma in situ without evidence of disease.
* History of leptomeningeal disease.
* Persons who have small cell carcinoma.
* Persons who do not meet the Stage IIIA NSCLC classification criteria outlined above.
* Presence of superior vena cava syndrome.
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 90 days after the last dose of trial treatment.
* Active central nervous system (CNS) metastases. Subjects must undergo a head computed tomography (CT) scan or brain MRI within 42 days prior to registration for protocol therapy to exclude brain metastases if symptomatic or without prior brain imaging.
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy.
* Patients should not have received any prior therapy for the current diagnosis of NSCLC. Treatments done for previously diagnosed malignancies are permitted. Prior therapy with a PD-1, PD-L1 (including Durvalumab), PD-L2 or CTLA-4 inhibitor or a lung cancer-specific vaccine therapy are not permitted.
* Presence of metastatic disease (stage IV NSCLC) is not allowed. Subjects must be evaluated with a CT or PET scan prior to registration for protocol therapy to exclude metastatic disease.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  * Patients with celiac disease controlled by diet alone
* Interstitial lung disease or history of pneumonitis requiring treatment with corticosteroids
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* History of psychiatric illness or social situations that would limit compliance with study requirements
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the investigator.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the investigator.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator.
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects with HIV/AIDS with adequate antiviral therapy to control viral load would be allowed. Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy. Testing not required.
* Has received a live vaccine within 30 days prior to planned start of study therapy. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* History of allograft or allogeneic bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg A Durm, MD, Principal Investigator — Indiana University School of Medicine
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon, Indianapolis, Indiana
  - New York University Clinical Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Neoadjuvant chemotherapy(Durvalumab, Paclitaxel, Carboplatin), radiation and immunotherapy (durvalumab) followed by surgical resection followed by adjuvant immunotherapy (durvalumab)
  Durvalumab: Neoadjuvant Durvalumab 750 mg IV on Days 1, 15 and 29
  Adjuvant Durvalumab 12 weeks after undergoing surgical resection 1,500 mg IV on Day 1
  Paclitaxel: Paclitaxel 45 mg/m2 IV Days 1, 8, 15, 22, 29 and +/- 36
  Carboplatin: Carboplatin AUC of 2 IV Days 1, 8, 15, 22, 29 +/- 36
  Radiation: 1.8-2.0 Gy per day (5 days/week) for a total of 45-61.2 Gy over 5-6 weeks. Treatment will be delivered using IMRT or 3DCRT using typically 6-10MV photons. Proton therapy is also allowed. 4D simulation and appropriate IGRT are encouraged. Radiation therapy must begin within one week of the first day of chemotherapy (or vice versa).
  Surgical Resection: Patients will undergo repeat imaging between 4 and 12 weeks after completing neoadjuvant therapy. Those without evidence of progressive disease and found to be a surgical candidate by a thoracic surgeon will undergo surgical resection between 4 and 12 weeks after neoadjuvant therapy.
Period: Overall Study
Arm/Group | Treatment
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 66 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
Baseline ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction, 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, and 5=Dead
  Participants
    ECOG = 0 | 3
    ECOG = 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: Pathologic Complete Response Rate is defined as lack of evidence of viable cancer in the surgical specimen at the time of surgery.
Time Frame: 3 months
Population: 4 Subjects completed the surgical procedure and were evaluable for Pathologic Complete Response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 4
Participants
  Pathological Complete Response Achieved | 0
  Pathological Complete Response Not Achieved | 4

2. Secondary Outcome: Pathologic N0 Rate
Description: Pathologic N0 rate is defined as a lack of evidence of viable cancer in the removed lymph nodes at the time of surgery.
Time Frame: 3 months
Population: 4 subjects completed the surgical procedure and were evaluable for Pathologic N0 status
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 4
Participants
  Pathologic N0 Status Achieved | 3
  Pathologic N0 Status Not Achieved | 1

3. Secondary Outcome: Assess Adverse Events (AE)
Description: Adverse events, >= grade 3 and related to treatment will be summarized by frequency and severity according to the NCI Common Terminology Criteria for (NCI CTCAE) v5
Time Frame: AEs had been recorded from time of signed informed consent until 90 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 13 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 6
Participants
  LUNG INFECTION Grade 5 | 1
  HYPOKALEMIA Grade 4 | 1
  ACIDOSIS Grade 3 | 1
  APPENDICITIS Grade 3 | 1
  PAIN Grade 3 | 1

4. Secondary Outcome: Disease Free Survival (DFS)
Description: Disease free survival will be defined as the time from surgical resection until the criteria for disease recurrence is met or death as a result of any cause. Disease recurrence is return of the cancer to where it started (local) or in another part of the body (distant).
Time Frame: Time from surgical resection until disease recurrence or death, up to a maximum of 8 months
Population: 4 patients out of 6 are evaluable for DFS. 2 patients did not go through the surgery and no response was recorded.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment
Number analyzed (Participants) | 4
Months | 6.7 [0.8 to NA] — Not enough participants achieved response to calculate upper 95% CI.

ADVERSE EVENTS:
Time Frame: Adverse events had been recorded from time of signed informed consent until 90 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 13 months.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
APPENDICITIS (Infections and infestations) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=6)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 2 (2)
ANXIETY (Psychiatric disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 4 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (6)
DERMATITIS RADIATION (Injury, poisoning and procedural complications) | 1 (3)
DIARRHEA (Gastrointestinal disorders) | 2 (2)
DIZZINESS (Nervous system disorders) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (3)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 4 (6)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 1 (1)
FATIGUE (General disorders) | 6 (7)
FEVER (General disorders) | 1 (4)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 2 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (4)
HYPOTENSION (Vascular disorders) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
INTRAOPERATIVE ARTERIAL INJURY (Injury, poisoning and procedural complications) | 1 (1)
LUNG INFECTION (Infections and infestations) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (8)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN (General disorders) | 2 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (2)
VOMITING (Gastrointestinal disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT03871153/Prot_SAP_000.pdf